CLINICAL TRIAL: NCT00895349
Title: The Impact of Positron Emission Tomography (PET) Imaging in Women With Locally Advanced Cervical Cancer
Brief Title: Impact of Positron Emission Tomography (PET) Imaging in Women With Locally Advanced Cervical Cancer (PET LACE Trial)
Acronym: PET LACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OCOG-2009-PETLACE
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancer; Squamous Cell Carcinoma; Adenosquamous Carcinoma; Adenocarcinoma
Keywords: Positron Emission Tomography (PET); Diagnostic Intervention; Locally Advanced Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma, Squamous Cell; Carcinoma, Adenosquamous; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CT Abdomen and Pelvis + whole body PET-CT
  Interventions: Procedure: CT Abdomen and Pelvis scan + whole body PET-CT scan
- 2 (Active Comparator): CT Abdomen and Pelvis
  Interventions: Procedure: CT Abdomen and Pelvis scan

INTERVENTIONS:
Procedure: CT Abdomen and Pelvis scan + whole body PET-CT scan — Pre-treatment scan
  Arms: 1
Procedure: CT Abdomen and Pelvis scan — Pre-treatment scan
  Arms: 2

SUMMARY:
The purpose of this trial is to improve the clinical management and outcome of patients with locally advanced cervical cancer by using positron emission tomography-computed tomography (PET-CT) imaging.

There is considerable debate worldwide regarding the utility of PET for staging cervical cancer. Although there are studies on the accuracy (sensitivity and specificity) of PET in cervical cancer, there are currently no prospective randomized studies on how PET information affects treatment decisions and outcomes.

DETAILED DESCRIPTION:
Cervical cancer is the second most common cause of cancer deaths worldwide. In Canada, it is estimated that in 2009 there will be 1,300 new cases of cervical cancer and that 380 women will die of this disease. The corresponding 2009 data for Ontario is 500 new cases and 140 deaths. In Canada, cervical cancer screening with the Pap test allows for the diagnosis and curative treatment of precancerous lesions of the cervix or early cervical cancers. Symptoms of cervical cancer include vaginal bleeding and discharge. Unfortunately these are often associated with more advanced disease.

The costs associated with health care are increasing. PET is an expensive imaging modality. Given that resources for health care are not unlimited, there needs to be high quality evidence of an intervention such as PET's efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women with newly diagnosed histologically confirmed FIGO Stage IB-IVA carcinoma of the cervix, including squamous, adenosquamous or adenocarcinoma. Women not suitable for surgery due to comorbidities (medical or other conditions) are also considered eligible.
* Age equal to or greater than 18 years
* Being considered for treatment with curative intent using concurrent chemotherapy and pelvic RT.

Exclusion Criteria:

* ECOG performance status greater than 2.
* Other cervical cancer tumour types (e.g. neuroendocrine, serous).
* Carcinoma of the cervical stump.
* Prior hysterectomy.
* Patients who, at the time of the initial evaluation, have already undergone a whole body PET-CT within the last 6 months.
* Contraindications to 18FDG PET-CT or CT of the abdomen and pelvis.
* Inability to lie supine for imaging with PET-CT.
* Contraindication to radiotherapy (i.e., significant Crohn's disease).
* Contraindication to cisplatin chemotherapy (i.e., non-reversible renal failure).
* Inadequate bone marrow function: ANC less than 1.5 X 10^9, platelets less than 100 X 10^9.
* Inadequate renal function: Creatinine greater/equal to 150 micromol/L
* Inadequate hepatic function: Bilirubin greater than 1.5 X ULN and SGOT and Alkaline Phosphatase greater than 3 X ULN.
* History of another invasive malignancy within the previous 5 years with the exception of non-melanoma skin cancer.
* Other medical conditions that may preclude chemo-radiation therapy.
* Known pregnancy or lactating.
* Inability to complete study or required follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Treatment delivered between patients having whole body 18FDG PET-CT in addition to CT of the abdomen and pelvis versus patients having a CT of the abdomen and pelvis alone. | 2 years

SECONDARY OUTCOMES:
Event free survival (EFS) of all patients. | 5 years
Overall Survival (OS) of all patients. | 5 years
Economic and Quality of Life analyses of all patients. | 2 years
Standardized Uptake Value (SUV) in predicting the EFS and OS of all patients. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Elit, MD, Principal Investigator — Juravinski Cancer Centre, Canada; Anthony Fyles, MD, Principal Investigator — Princess Margaret Hospital, Canada; Greg Pond, PhD, Principal Investigator — Ontario Clinical Oncology Group/McMaster University, Department of Oncology; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group/McMaster University, Department of Oncology; Karen Gulenchyn, MD, Principal Investigator — Hamilton Health Sciences Centre; Mostafa Atri, MD, Principal Investigator — University Health Network, Toronto; Douglas Coyle, PhD, Principal Investigator — University of Ottawa Epidemiology & Community Medicine
Locations (6):
- Canada (6):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Odette Cancer Centre (Toronto-Sunnybrook), Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Elit LM, Fyles AW, Gu CS, Pond GR, D'Souza D, Samant R, Anthes M, Thomas G, Filion M, Arsenault J, Dayes I, Whelan TJ, Gulenchyn KY, Metser U, Dhamanaskar K, Levine MN. Effect of Positron Emission Tomography Imaging in Women With Locally Advanced Cervical Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2018 Sep 7;1(5):e182081. doi: 10.1001/jamanetworkopen.2018.2081. PMID 30646153